CLINICAL TRIAL: NCT00077441
Title: Phase II Trial of PS-341 in Patients With Hepatocellular Carcinoma
Brief Title: Bortezomib in Treating Patients With Hepatocellular Carcinoma (Liver Cancer)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02806; MC0255; N01CM62205 (NIH)
Record Dates: First submitted 2004-02-10; First posted 2004-02-12 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Adult Primary Hepatocellular Carcinoma; Advanced Adult Primary Liver Cancer; Localized Unresectable Adult Primary Liver Cancer; Recurrent Adult Primary Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Bortezomib

ARMS (1):
- Treatment (bortezomib) (Experimental): Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: bortezomib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well bortezomib works in treating patients with hepatocellular carcinoma (liver cancer) that cannot be removed with surgery. Bortezomib may stop the growth of tumor cells by blocking the enzymes necessary for their growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Proportion of confirmed tumor responses.

SECONDARY OBJECTIVES:

I. To evaluate the confirmed and objective response rate. II. To assess patient outcome as estimated by duration of response, time to disease progression, and survival.

III. To evaluate the adverse event rates associated with PS-341 in this population.

IV. To explore the relationships between laboratory correlates (eg. IHC) and patient outcome (eg p53 and disease progression).

V. To evaluate alterations in laboratory correlates from pre-treatment measurements (ie, pre and post treatment). The following immunohistochemistry (IHC) assays will be performed: IHC of p53, IHC of p21, IHC of p27, IHC of NFkB, IHC of Ki67.

OUTLINE: This is a multicenter study.

Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months until disease progression and then every 6 months for up to 3 years from study entry.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed hepatocellular carcinoma (HCC) that is not amenable to surgical resection
* Must have measurable disease; NOTE: For patients having only lesions measuring > 1 cm to =< 2 cm must use spiral CT imaging for all tumor assessments
* Absolute neutrophil count (ANC) >= 1500/mm^3
* PLT >= 75,000/mm^3
* Total bilirubin =< 3 x upper normal limit (UNL)
* Serum AST =< 5 x UNL
* Serum ALT =< 5 x UNL
* Serum creatinine =< 2 mg/dL
* Serum albumin >= 2.5 g/dL
* PT/ INR =< 1.5 (EXCEPTION - Patients with full-dose anticoagulants are eligible provided the patient has been on a stable dose, >= 2 weeks, of warfarin or low molecular weight heparin and has an PT/INR range 2-3)
* Child-Pugh classification of A or B
* Patients may not have received prior systemic chemotherapy BUT may have received prior chemoembolization, cryotherapy, radiofrequency ablation, ethanol injection, or photodynamic therapy, provided the following criteria are met:

  * > 6 weeks has elapsed since that therapy
  * Indicator lesion(s) is/are outside the area of prior treatment or, if the only indicator lesion is inside the prior treatment area, there must be clear evidence of disease progression associated with that lesion
  * Edges of the indicator lesion are clearly distinct on CT scanning
* ECOG performance status (PS) 0, 1, or 2
* Estimated life expectancy >= 24 weeks
* Capable of understanding the investigational nature, potential risks and benefits of the study and able to provide written informed consent

Exclusion Criteria:

* Any of the following:

  * Prior systemic anticancer therapy. Note: Chemoembolization is allowed and for trial purposes is not considered a systemic chemotherapy; however, >= 6 weeks must have elapsed between chemoembolization and enrollment on this study
  * Prior PS-341 therapy
  * Immunotherapy =< 4 weeks have elapsed prior to study entry
  * Biologic therapy =< 4 weeks have elapsed prior to study entry
  * Radiation therapy =< 4 weeks have elapsed prior to study entry
  * Cryotherapy =< 6 weeks have elapsed since prior to study entry
  * Radiofrequency ablation =< 6 weeks have elapsed since prior to study entry
  * Ethanol injection =< 6 weeks have elapsed since prior to study entry
  * Photodynamic therapy =< 6 weeks have elapsed since prior to study entry
  * Major surgery, or significant traumatic injury =< 3 weeks prior to study entry
  * Other concurrent chemotherapy, immunotherapy, radiotherapy, or any other therapy or supportive care considered investigational
* Presence of > grade 1 sensory peripheral neuropathy of any etiology OR grade 1 with neuropathic pain of any etiology
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to PS-341
* History of other malignancy =< 3 years prior to study entry, except for adequately treated basal cell or squamous cell skin cancer
* Any of the following as this regimen may be harmful to a developing fetus or nursing child:

  * Pregnant women
  * Breastfeeding women
  * Men or women of childbearing potential or their sexual partners who are unwilling to employ adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, or abstinence, etc.)
* Known CNS metastases
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris, cardiac arrhythmia
  * Psychiatric illness that would limit compliance with study requirements
* HIV-positive patients receiving combination anti-retroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2005-04; Primary Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Proportion of confirmed tumor responses, defined to be either a CR or PR noted as the objective status on 2 consecutive evaluations at least 6 weeks apart | Up to 36 weeks (12 courses)
  Ninety-five percent confidence intervals for the true success proportion will be calculated.

SECONDARY OUTCOMES:
Survival time | Time from registration to death due to any cause, assessed up to 3 years
  The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time to disease progression | Time from registration to documentation of disease progression, assessed up to 3 years
  The distribution of time to progression will be estimated using the method of Kaplan-Meier.
Duration of response is defined for all evaluable patients who have achieved an objective response as the date at which the patient's objective status is first noted to be either a CR or PR to the date progression is documented | Up to 3 years
Time to treatment failure | Time from the date of registration to the date at which the patient is removed from treatment due to progression, toxicity, or refusal, assessed up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: George Kim, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States